CLINICAL TRIAL: NCT00919711
Title: A Randomized Open-Label Study to Evaluate the Safety and Efficacy of Denosumab and Monthly Actonel® Therapies in Postmenopausal Women Transitioned From Weekly or Daily Alendronate Therapy
Brief Title: Study to Evaluate the Safety and Efficacy of Denosumab and Actonel® in Post Menopausal Women Transitioned From Alendronate Therapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20080099
Record Dates: First submitted 2009-06-11; First posted 2009-06-12 (Estimated); Results first posted 2012-12-12 (Estimated); Last update posted 2020-07-28 (Actual); Status verified 2020-03

CONDITIONS: Osteoporosis
Keywords: Menopausal Osteoporosis
MeSH Terms: conditions — Osteoporosis; Osteoporosis, Postmenopausal | interventions — Risedronic Acid; Denosumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Denosumab 60 mg (Experimental)
  Interventions: Drug: Denosumab
- Risedronate 150 mg QM (Active Comparator)
  Interventions: Drug: Actonel®

INTERVENTIONS:
Drug: Actonel® — Oral Actonel® (Risedronate) in total a 150mg per month (one 75mg tablet to be taken on each of 2 consecutive days per month).
  Other Names: Risedronate
  Arms: Risedronate 150 mg QM
Drug: Denosumab — Denosumab 60 mg, once every 6 months, Subcutaneous
  Arms: Denosumab 60 mg

SUMMARY:
A randomized, open label study to assess the safety and effectiveness of Denosumab, administered every 6 months and Actonel ® (Risedronate), administered monthly in post menopausal women transitioned from weekly or daily Alendronate therapy.

ELIGIBILITY:
Inclusion Criteria:

* Ambulatory, post menopausal women aged 55 years or older at screening. Have received their first prescription of daily or weekly alendronate therapy, for the treatment for post menopausal osteoporosis at least 1 month prior to screening. Use of raloxifene, calcitonin or hormone replacement therapy (HRT) prior to alendronate treatment will be allowed. Prior and/or current use of vitamin D and calcium will be allowed.
* Has stopped oral alendronate therapy (is denoted as non-persistent) before the screening visit or, is still taking oral alendronate therapy but does not take on a regular basis (this will be assessed by the completion of a compliance questionnaire at screening).
* Provide signed informed consent before any study-specific procedures are conducted.

Exclusion Criteria:

* Any prior or current use of medications prescribed for osteoporosis treatment other than oral daily alendronate, calcium and vitamin D. Prior use of raloxifen, calcitonin or HRT before alendronate therapy was started will be allowed.
* Hypersensitivity to Actonel® or any ingredient of Actonel® tablets.
* Contraindicated or poorly tolerant of alendronate therapy.
* Active gastric or duodenal ulcer.
* Known sensitivity to mammalian cell derived products.
* Known intolerance to calcium supplements.
* Malignancy within the last 5 years (except for cervical or basal cell carcinoma).
* Vitamin D deficiency (serum 25-OH vitamin D less than 20ng/mL (equivalent to 49.9 nanomoles per Liter) at screening.
* Current hypo- or hypercalcemia based on the central laboratory reference ranges.
* Uncontrolled hyper- or hypothyroidism (stable on antithyroid therapy or post-ablation is allowed, if the laboratory results from screening show that thyroid stimulating hormone (TSH) is within the normal range).
* Any metabolic bone disease, e.g., osteomalacia or osteogenesis imperfecta, Paget's disease of bone that may interfere with the interpretation of the findings.
* Height, weight or girth which may preclude accurate dual x-ray absorptiometry (DXA measurements).
* Fewer than 2 lumbar vertebrae (L1-L4) able to be evaluated by DXA.
* Known to have tested positive for human immunodeficiency virus.
* Previous participation in clinical trials with denosumab within the last 12 months (regardless of treatment).
* Any laboratory abnormality, physical or psychiatric disorder (including substance abuse in last 12 months) which, in the opinion of the investigator, will prevent the subject from giving written informed consent or completing the study or interfere with the interpretation of the study results.
* Currently enrolled in or within 30 days of ending another investigational device or drug trial(s).

Min Age: 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 870 (Actual)
Dates: Start 2009-09-01 (Actual); Primary Completion 2011-12-21 (Actual); Study Completion 2012-03-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- [Background] Roux C, Hofbauer LC, Ho PR, Wark JD, Zillikens MC, Fahrleitner-Pammer A, Hawkins F, Micaelo M, Minisola S, Papaioannou N, Stone M, Ferreira I, Siddhanti S, Wagman RB, Brown JP. Denosumab compared with risedronate in postmenopausal women suboptimally adherent to alendronate therapy: efficacy and safety results from a randomized open-label study. Bone. 2014 Jan;58:48-54. doi: 10.1016/j.bone.2013.10.006. Epub 2013 Oct 17. PMID 24141036
- [Derived] Miller PD, Pannacciulli N, Malouf-Sierra J, Singer A, Czerwinski E, Bone HG, Wang C, Huang S, Chines A, Lems W, Brown JP. Efficacy and safety of denosumab vs. bisphosphonates in postmenopausal women previously treated with oral bisphosphonates. Osteoporos Int. 2020 Jan;31(1):181-191. doi: 10.1007/s00198-019-05233-x. Epub 2019 Nov 28. PMID 31776637
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled from 19 October 2009 through 4 January 2011
Groups:
- Risedronate 150 mg QM: Risedronate 150 mg oral once monthly
- Denosumab 60 mg Q6M: Denosumab 60 mg subcutaneous once every 6 months
Period: Overall Study
Arm/Group | Risedronate 150 mg QM | Denosumab 60 mg Q6M
Started | 435 | 435
Completed | 402 | 422
Not Completed | 33 | 13
Not completed — Withdrawal by Subject | 15 | 7
Not completed — Adverse Event | 13 | 3
Not completed — Other | 1 | 2
Not completed — Administrative Decision | 0 | 1
Not completed — Lost to Follow-up | 2 | 0
Not completed — Death | 1 | 0
Not completed — Noncompliance | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Risedronate 150 mg QM | Denosumab 60 mg Q6M | Total
Number analyzed (Participants) | 435 | 435 | 870
Age, Continuous [Mean (Standard Deviation); unit: Years] | 67.7 (6.8) | 67.8 (7.0) | 67.7 (6.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 435 | 435 | 870
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: Participants]
  White or Caucasian | 425 | 424 | 849
  Hispanic or Latino | 6 | 7 | 13
  Asian | 4 | 3 | 7
  Japanese | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Total Hip BMD Percent Change From Baseline at Month 12
Description: Bone Mineral Density Assessed by Dual Energy X-Ray Absorptiometry
Time Frame: Baseline to month 12
Population: All randomized subjects excluding those with missing post baseline data and missing covariate for regression imputation
Measure: Mean (95% Confidence Interval); unit: Percent Change From Baseline
Arm/Group | Risedronate 150 mg QM | Denosumab 60 mg Q6M
Number analyzed (Participants) | 434 | 432
Percent Change From Baseline | 0.5 [0.2 to 0.7] | 2.0 [1.8 to 2.3]
Statistical Analysis 1: Comparison: Risedronate 150 mg QM vs Denosumab 60 mg Q6M; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Net) = 1.6, 95% CI 2-sided [1.2 to 2.0] — Denosumab - Risedronate

2. Secondary Outcome: Serum CTX Percent Change From Baseline at Month 1
Description: Serum Type-1 Collagen C-Telopeptide Percent Change From Baseline at Month 1
Time Frame: Baseline to month 1
Population: All randomized subjects who enrolled in the bone marker substudy with observed data
Measure: Median (Inter-Quartile Range); unit: Percent Change From Baseline
Arm/Group | Risedronate 150 mg QM | Denosumab 60 mg Q6M
Number analyzed (Participants) | 68 | 84
Percent Change From Baseline | -17.0 [-36.8 to -1.6] | -77.7 [-85.9 to -67.6]
Statistical Analysis 1: Comparison: Risedronate 150 mg QM vs Denosumab 60 mg Q6M; Test type: Superiority or Other; p < 0.0001, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Femoral Neck BMD Percent Change From Baseline at Month 12
Description: Bone Mineral Density Assessed by Dual Energy X-Ray Absorptiometry
Time Frame: Baseline to month 12
Population: All randomized subjects excluding those with missing post baseline data and missing covariate for regression imputation
Measure: Mean (95% Confidence Interval); unit: Percent Change From Baseline
Arm/Group | Risedronate 150 mg QM | Denosumab 60 mg Q6M
Number analyzed (Participants) | 434 | 432
Percent Change From Baseline | 0.0 [-0.4 to 0.3] | 1.4 [1.0 to 1.7]
Statistical Analysis 1: Comparison: Risedronate 150 mg QM vs Denosumab 60 mg Q6M; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Net) = 1.4, 95% CI 2-sided [0.9 to 1.8] — Denosumab - Risedronate

4. Secondary Outcome: Lumbar Spine BMD Percent Change From Baseline at Month 12
Description: Bone Mineral Density Assessed by Dual Energy X-Ray Absorptiometry
Time Frame: Baseline to month 12
Population: All randomized subjects excluding those with missing post baseline data and missing covariate for regression imputation
Measure: Mean (95% Confidence Interval); unit: Percent Change From Baseline
Arm/Group | Risedronate 150 mg QM | Denosumab 60 mg Q6M
Number analyzed (Participants) | 434 | 432
Percent Change From Baseline | 1.1 [0.7 to 1.5] | 3.4 [3.1 to 3.8]
Statistical Analysis 1: Comparison: Risedronate 150 mg QM vs Denosumab 60 mg Q6M; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Net) = 2.3, 95% CI 2-sided [1.8 to 2.8] — Denosumab - Risedronate

ADVERSE EVENTS:
Time Frame: 12 months
Description: The table of Other Adverse Events summarizes the most frequent non-serious occurrences of adverse events.
Arm/Group | Risedronate 150 mg QM | Denosumab 60 mg Q6M
Serious Adverse Events (participants affected / at risk) | 35/429 | 33/429
Other Adverse Events (participants affected / at risk) | 0/429 | 0/429
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Risedronate 150 mg QM (N=429) | Denosumab 60 mg Q6M (N=429)
Atrial fibrillation (Cardiac disorders) | 0 | 2
Atrial flutter (Cardiac disorders) | 1 | 0
Cardiac arrest (Cardiac disorders) | 1 | 0
Coronary artery disease (Cardiac disorders) | 1 | 0
Coronary artery stenosis (Cardiac disorders) | 2 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0
Ventricular extrasystoles (Cardiac disorders) | 0 | 1
Talipes (Congenital, familial and genetic disorders) | 0 | 1
Macular hole (Eye disorders) | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0
Coeliac disease (Gastrointestinal disorders) | 0 | 1
Colonic pseudo-obstruction (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Diverticular perforation (Gastrointestinal disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 1
Malaise (General disorders) | 0 | 1
Bile duct stone (Hepatobiliary disorders) | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 1
Jaundice (Hepatobiliary disorders) | 0 | 1
Anaphylactic shock (Immune system disorders) | 1 | 0
Appendicitis (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 1 | 0
Diverticulitis (Infections and infestations) | 0 | 1
Herpes zoster (Infections and infestations) | 1 | 0
Intervertebral discitis (Infections and infestations) | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0
Pneumonia chlamydial (Infections and infestations) | 1 | 0
Respiratory tract infection (Infections and infestations) | 0 | 1
Sinusitis (Infections and infestations) | 0 | 1
Urosepsis (Infections and infestations) | 0 | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 | 1
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1
Fibula fracture (Injury, poisoning and procedural complications) | 0 | 1
Foot fracture (Injury, poisoning and procedural complications) | 1 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 0
Joint injury (Injury, poisoning and procedural complications) | 1 | 0
Lip injury (Injury, poisoning and procedural complications) | 1 | 0
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1
Procedural pain (Injury, poisoning and procedural complications) | 0 | 1
Pubis fracture (Injury, poisoning and procedural complications) | 0 | 1
Radius fracture (Injury, poisoning and procedural complications) | 0 | 2
Ulna fracture (Injury, poisoning and procedural complications) | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 2
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1
Meniscal degeneration (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 2
Anal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to neck (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Carotid artery occlusion (Nervous system disorders) | 0 | 1
Carotid artery stenosis (Nervous system disorders) | 1 | 0
Carpal tunnel syndrome (Nervous system disorders) | 1 | 0
Cerebral ischaemia (Nervous system disorders) | 0 | 2
Cerebrovascular accident (Nervous system disorders) | 0 | 2
Presyncope (Nervous system disorders) | 1 | 0
Radicular syndrome (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 0 | 1
Haematuria (Renal and urinary disorders) | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 1
Vaginal prolapse (Reproductive system and breast disorders) | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Bronchopneumopathy (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Phlebitis (Vascular disorders) | 1 | 0
Temporal arteritis (Vascular disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results aftercompletion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.